CLINICAL TRIAL: NCT06428097
Title: Levothyroxine Supplementation for Heart Transplant Recipients: A Randomized Control Trial
Brief Title: Levothyroxine Supplementation for Heart Transplant Recipients
Acronym: Levo
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-39323
Record Dates: First submitted 2024-05-03; First posted 2024-05-24 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Heart Transplant Failure; Heart Transplant Infection
MeSH Terms: interventions — Thyroxine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Levothyroxine (Experimental): Patients will be double-blinded and randomized to receive levothyroxine.
  Interventions: Drug: Levothyroxine
- No Levothyroxine (Placebo Comparator): Patients will be double-blinded and randomized to receive no levothyroxine. The placebo will be normal saline.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Levothyroxine — Dosing will be based on pre-existing protocols in the setting of organ donation.This will be the protocol for the first 18-38 hours starting intra-operatively after the donated heart is sewn in.
  Arms: Levothyroxine
Drug: Normal saline — Placebo will be normal saline and will be dosed at the same rate and time as the study drug.
  Arms: No Levothyroxine

SUMMARY:
This will be a prospective, randomized study performed at a single tertiary referral academic medical center (University of California San Francisco, CA), evaluating the survival benefits of levothyroxine compared with no levothyroxine for patients who have undergone heart transplant. It will be double-blinded and placebo-control; participants will be randomized to receive levothyroxine or receive no levothyroxine.

DETAILED DESCRIPTION:
Studies have shown that thyroid hormone results in a higher number of organs available for transplant. Increasingly, thyroid hormone supplementation is used amongst transplant donors. However, it is not the current standard of practice to supplement recipients without a prior medical history of hypothyroidism with levothyroxine. Two large retrospective studies have demonstrated improved 30-days survival and lower risk of all-cause mortality for heart transplant recipients who receive levothyroxine in the post-operative context. No randomized trials have tested this hypothesis and so the investigators aim to trial the use of levothyroxine for heart transplant recipients at University of California San Francisco using a double-blinded and placebo controlled randomized control trial study design. This will be a prospective, randomized study performed at a single tertiary referral academic medical center (University of California San Francisco, CA), evaluating the survival benefits of levothyroxine compared with no levothyroxine for patients who have undergone heart transplant. It will be double-blinded and placebo-control; participants will be randomized to receive levothyroxine or receive no levothyroxine.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be listed for heart transplantation
2. Age ≥18 years
3. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with pre-existing thyroid related condition including hypothyroidism, hyperthyroidism and malignancy
2. Patients with a known allergy or intolerance to levothyroxine
3. Patients participating in another study evaluating an investigational drug within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who receive Levothyroxine's vasopressor use compared to number of participants who receive normal saline's vasopressor use. | 35 months total completion, 18 months accrual, 12 months follow up and 5 months data analysis
  Measured using the vasoactive-inotropic score (VIS) scale.
  VIS calculation: dopamine dose (μg/kg/min) + dobutamine dose (μg/kg/min) + 100 × epinephrine dose (μg/kg/min) + 10 × milrinone dose (μg/kg/min) + 10 000 × vasopressin dose (unit/kg/min) + 100 × norepinephrine dose (μg/kg/min)

SECONDARY OUTCOMES:
Do the participants receiving levothyroxine experience lower frequencies of primary graft dysfunction? | 35 months total completion, 18 months accrual, 12 months follow up and 5 months data analysis
  Measured as a yes or no diagnosis.
Does the total vasoactive-inotropic score (VIS) decrease for patients who receive levothyroxine? | 35 months total completion, 18 months accrual, 12 months follow up and 5 months data analysis
  Measured using the vasoactive-inotropic score (VIS) scale.
  VIS calculation: dopamine dose (μg/kg/min) + dobutamine dose (μg/kg/min) + 100 × epinephrine dose (μg/kg/min) + 10 × milrinone dose (μg/kg/min) + 10 000 × vasopressin dose (unit/kg/min) + 100 × norepinephrine dose (μg/kg/min)
Do the participants have improved cardiac output? | 35 months total completion, 18 months accrual, 12 months follow up and 5 months data analysis
  Cardiac output is calculated using stroke volume and heart rate and measured in liters/minute.
  (Cardiac output = stroke volume x heart rate)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Smith, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes